CLINICAL TRIAL: NCT01663324
Title: Repetitive Transcranial Magnetic Stimulation for the Treatment of Chronic Tinnitus: Optimization by Stimulation of the Cortical Tinnitus Network
Brief Title: rTMS for the Treatment of Chronic Tinnitus: Optimization by Simulation of the Cortical Tinnitus Network
Acronym: Multisite rTMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Berthold Langguth, MD, Ph.D., MD, Ph.D., University of Regensburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Uni-Reg-multisite-rTMS-Tin-01
Record Dates: First submitted 2012-07-23; First posted 2012-08-13 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Tinnitus
Keywords: Tinnitus; chronic subjective Tinnitus; transcranial magnetic stimulation; rTMS; hearing disorders
MeSH Terms: conditions — Tinnitus; Hearing Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- single site rTMS (Experimental): Low frequency temporoparietal transcranial magnetic stimulation
  Intervention: Device: rTMS intervention 1
  Interventions: Device: rTMS intervention 1
- multisite rTMS (Experimental): Combined high frequency dorsolateral prefrontal (unilateral) and low frequency temporoparietal (bilateral) stimulation
  Intervention: Device: rTMS Intervention 2
  Interventions: Device: rTMS intervention 2

INTERVENTIONS:
Device: rTMS intervention 1 — Low frequency rTMS (Magventure Mag Pro Option) applied over left temporoparietal cortex: 3000 stimuli of 1Hz rTMS (110% motor threshold); 1 minute break after 1000 and 2000 stimuli.
  Arms: single site rTMS
  Arms: single site rTMS
Device: rTMS intervention 2 — Repetitive transcranial magnetic stimulation (Magventure Mag Pro Option): 1000 stimuli of 20 Hz rTMS over the left DLPFC (110% motor threshold) followed by 1000 stimuli of 1 Hz rTMS over the left temporoparietal cortex (110% motor threshold) followed by 1000 stimuli of 1 Hz rTMS over right temporoparietal cortex (110% motor threshold).
  Arms: multisite rTMS
  Arms: multisite rTMS

SUMMARY:
Transcranial Magnetic Stimulation is used to modulate both the auditory and non-auditory neural pathways contributing to the perception of phantom sounds.

DETAILED DESCRIPTION:
Tinnitus is the phantom auditory perception of sound in the absence of an external or internal acoustic stimulus. It is a frequent problem which can interfere significantly with the ability to lead a normal life. Treatment remains difficult. Most available therapies focus on habituation rather than treating the cause. Tinnitus has been shown to be associated with functional reorganization of auditory neural pathways and tonotopic maps in the central auditory system. Consequently, low-frequency Repetitive Transcranial Magnetic Stimulation (rTMS) applied to the temporoparietal areas has been investigated for the treatment of tinnitus. Additionally, there is growing evidence that a neural network of both auditory and non-auditory cortical areas is involved in the pathophysiology of chronic subjective tinnitus. Targeting several core regions of this network by rTMS might constitute a promising strategy to enhance treatment effects. A new multisite treatment protocol which is supposed to have an effect on both auditory and non-auditory cortical areas will be examined with regard to feasibility, safety and clinical efficacy in patients suffering from chronic tinnitus in a controlled pilot trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of subjective chronic tinnitus
* THI > 38
* Duration of tinnitus more than 6 months

Exclusion Criteria:

* Objective tinnitus
* Treatable cause of the tinnitus
* Involvement in other treatments for tinnitus at the same time
* Clinically relevant psychiatric comorbidity
* Clinically relevant unstable internal or neurological comorbidity
* History of or evidence of significant brain malformation or neoplasm, head injury
* Cerebral vascular events
* Neurodegenerative disorder affecting the brain or prior brain surgery;
* Metal objects in and around body that can not be removed
* Pregnancy
* Alcohol or drug abuse
* Prior treatment with TMS

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-07; Primary Completion 2014-08 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Number of treatment responders (TQ reduction ≥5, contrast baseline versus day 12) | Day 12
Change of tinnitus severity as measured by the Tinnitus Questionnaire of Goebel&Hiller (contrast baseline versus day 12) | Day 12

SECONDARY OUTCOMES:
Change of depressive symptoms as measured by the Major Depression Inventory (MDI) | Day 12
Change in quality of life as measured by the WHOQoL | Day 12
Change in hyperacusis as measured by the German questionnaire "Geräuschüberempfindlichkeitsfragebogen" | Day 12
Number of treatment responders (TQ reduction ≥5, contrast Baseline versus day 90) | Day 90
Change of tinnitus severity as measured by the Tinnitus Handicap Inventory (THI) and Tinnitus Severity Scale | Day 12
Change of tinnitus severity as measured by the Tinnitus Handicap Inventory (THI) and Tinnitus Severity Scale | Day 90
Change of tinnitus severity as measured by the Tinnitus Handicap Inventory (THI) and Tinnitus Severity Scale | Day 180
Change of depressive symptoms as measured by the Major Depression Inventory (MDI) | Day 180
Change of depressive symptoms as measured by the Major Depression Inventory (MDI) | Day 90
Change in quality of life as measured by the WHOQoL | Day 90
Change in quality of life as measured by the WHOQoL | Day 180
Change in hyperacusis as measured by the German questionnaire "Geräuschüberempfindlichkeitsfragebogen" | Day 90
Change in hyperacusis as measured by the German questionnaire "Geräuschüberempfindlichkeitsfragebogen" | Day 180
Number of treatment responders (TQ reduction ≥5, contrast Baseline versus day 180) | Day 180
Change of tinnitus severity as measured by the Tinnitus Questionaire of Goebel&Hiller | Day 90
Change of tinnitus severity as measured by the Tinnitus Questionaire of Goebel&Hiller | Day 180

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Langguth, MD, Ph.D., Principal Investigator — University of Regensburg, Dept of Psychiatry
Locations (1):
- University of Regensburg- Dept of Psychiatry, Regensburg, Germany

REFERENCES:
- [Result] Lehner A, Schecklmann M, Greenlee MW, Rupprecht R, Langguth B. Triple-site rTMS for the treatment of chronic tinnitus: a randomized controlled trial. Sci Rep. 2016 Mar 1;6:22302. doi: 10.1038/srep22302. PMID 26927363
- [Derived] Lehner A, Schecklmann M, Kreuzer PM, Poeppl TB, Rupprecht R, Langguth B. Comparing single-site with multisite rTMS for the treatment of chronic tinnitus - clinical effects and neuroscientific insights: study protocol for a randomized controlled trial. Trials. 2013 Aug 23;14:269. doi: 10.1186/1745-6215-14-269. PMID 23968498